CLINICAL TRIAL: NCT00504478
Title: Effect of HCCD Supplemented With Omega-3 Fatty-Acids on Inflammation in Healthy, Overweight Subjects
Acronym: HCCD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TASMC-07-BS-164-CTIL
Record Dates: First submitted 2007-07-19; First posted 2007-07-20 (Estimated); Last update posted 2007-07-20 (Estimated); Status verified 2007-04

CONDITIONS: Inflammation
Keywords: Inflammation; carbohydrates; omega-3; overweight; diet
MeSH Terms: conditions — Inflammation; Overweight | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 8-weeks of high complex carbohydrate diet
  Interventions: Other: high complex carbohydrate diet
- 2 (Experimental): omega-3 fatty acids supplements
  Interventions: Dietary Supplement: omega-3 fatty acids; Other: high complex carbohydrate diet

INTERVENTIONS:
Dietary Supplement: omega-3 fatty acids — omega-3 supplement will be given in addition to high complex carbohydrate diet.
  Arms: 2
Other: high complex carbohydrate diet

SUMMARY:
The purpose of this study is to examine the anti inflammatory effect of high complex carbohydrate diet, supplemented by omega-3 fatty acids.

DETAILED DESCRIPTION:
Background: Atherosclerosis is the main cause for premature morbidity and mortality in the western world. It becomes evident that one of the main causes for development of atherosclerosis is the presence of low grade, internal inflammation. The inflammatory process leads to endothelial dysfunction, the early event in the pathogenesis of atherosclerosis. The inflammatory process is known to be induced by several factors such as obesity, recurring infections, smoking, and sedentary lifestyle. It was found that weight reduction decreased sub clinical inflammation. It was also found that the composition of the diet affects the inflammatory process.

Working hypothesis and aims: Our preliminary results show that high complex carbohydrate diet (HCCD) has beneficial effect on several markers of inflammation. The aims of this study are to reinforce our preliminary results by measuring the effect of HCCD on additional markers of inflammation (TNFα, IL6) and of endothelial dysfunction (ICAM-1, VCAM-1), and to identify the genes affected by HCCD in monocytes. In addition the aim of this study is to determine whether consumption of omega-3 oil actually increase the anti-inflammatory effect obtained by HCCD.

Methods: 150 healthy overweight volunteers will be divided into 2 groups; HCCD group and HCCD supplemented with the omega-3 fatty acids. Blood sample will be taken following an overnight 12 hour fast, before and after 8 weeks diet, for the following analysis: total cell count, plasma lipids, glucose and insulin, erythrocyte sedimentation rate, fibrinogen, white blood cell count, and CRP. Markers of leukocyte activation will be determined using FACS analysis. In addition, using ELISA, the following pro and anti inflammatory cytokines and markers for endothelial dysfunction will be analyzed: VCAM-1 and ICAM-1. Micro array analysis for genes transcription differences induced by HCCD will be performed in monocytes using Affymetrix chips.

Expected results: We assume that HCCD consumption may improve the inflammatory markers as well as markers of endothelial dysfunction and affect expression of genes involved in inflammation in monocytes. In addition we assume that omega-3 fatty acids will strengthen the positive effect of HCCD on parameters of inflammation.

Importance and probable implications to Medicine: The results of this study may establish scientific basis for guiding people for healthy lifestyle, including the consumption of diet composed of components with anti inflammatory effects, as well as nutritional supplements enhancing anti-inflammatory properties of the diet. This work will also be able to establish the influence of the diet and supplementations on gene expression for inflammatory reaction in monocytes.

ELIGIBILITY:
Inclusion Criteria:

* 150 healthy overweight volunteers

Exclusion Criteria:

* Individuals who had an infective/inflammatory disease during the six month period prior to the commencement of the study, and individuals who are on treatment with statins or any steroidal or non steroidal anti inflammatory agents, except for aspirin at a dose of up to 325 mg/day, will be excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2008-01; Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
markers of inflammation | 2 years

SECONDARY OUTCOMES:
difference in the pattern of monocyte gene expression | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Shlomo Berliner, MD PhD, Principal Investigator — The Tel Aviv Sauraski Medical Center